CLINICAL TRIAL: NCT05885906
Title: Aloe Vera Versus Thyme Honey Mouthwash in Management of Xerostomia in Type 2 Diabetics (A Randomized Controlled Clinical Trial With Biochemical Analysis)
Brief Title: Aloe Vera Versus Thyme Honey Mouthwash in Management of Xerostomia in Type 2 Diabetics
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dina Borham Abdelhafez Abdellatif Elkhouly, Resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FDASU-RecIM122208
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Xerostomia
Keywords: Xerostomia; Aloevera; Thyme honey; type 2 diabetes
MeSH Terms: conditions — Xerostomia; Diabetes Mellitus, Type 2 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aloevera group (Active Comparator): 15 patients suffering from diabetes induced xerostomia that will receive aloe vera as mouthwash (20 ml of aloe vera 50%) 3 times per day for 4 weeks.
  Interventions: Drug: Aloevera
- Thyme honey group (Active Comparator): 15 patients suffering from diabetes induced xerostomia that will receive thyme honey mouthwash (20 ml of thyme honey diluted in 100 ml of distilled water) 3 times per day for 4 weeks.
  Interventions: Drug: Thyme honey
- Saline group (Placebo Comparator): 15 patients suffering from diabetes induced xerostomia that will receive saline mouthwash as a control group (20 ml of saline) 3 times per day for 4 weeks.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Aloevera — Mouthwash
  Arms: Aloevera group
Drug: Thyme honey — Mouthwash
  Arms: Thyme honey group
Drug: Saline — Mouthwash
  Arms: Saline group

SUMMARY:
The objectives of the present study are to:

1. Compare the clinical efficacy of (50%) aloe vera versus (20%) thyme honey mouthwash on management of xerostomia in diabetic patients by measuring the salivary flow rate as a primary objective.
2. Asses the biochemical effect of aloe vera and thyme honey on the level of salivary nitric oxide, xerostomia grade as well as patient quality of life as a secondary objective.

Research question:

Which is better aloe vera or thyme honey in improving salivary flow rate in diabetic patients suffering from xerostomia?

Patient Grouping and Randomization:

Patients with xerostomia will be randomly distributed into three groups using a computer-generated randomization table. Allocation concealment will be achieved by a sealed opaque envelope with a ratio of 1:1:1

Group 1 (Aloe Vera group)

Include (15) patient suffering from diabetes induced xerostomia that will receive aloe vera as mouthwash

Group 2 (Thyme honey group):

Include (15) patient suffering from diabetes induced xerostomia that will receive thyme honey mouthwash

Group 3 (Saline control group):

Include (15) patient suffering from diabetes induced xerostomia that will receive saline mouthwash

DETAILED DESCRIPTION:
Saliva is a complex mix from major as well as minor salivary glands and gingival crevicular fluids. It is a clear and slightly acidic diluted secretion with more than 99% water, electrolytes, immunoglobulins, enzymes, proteins, mucin and nitrogenous products. Subjective feeling of a dry mouth is known as xerostomia, which may result from diminished saliva production, but some people reported feeling a dry mouth even though there was no decrease in saliva quantity.Diabetes mellitus is considered one of the main causes of xerostomia There are different treatments modalities of xerostomia which include pharmacological and non-pharmacological treatments.Recently different herbs were used in the treatment of xerostomia and showed promising results and great patient acceptance among which aloe vera and thyme honey are used.

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, with type 2 diabetes mellitus only and suffering from xerostomia.
2. Patients willing to follow all the instructions and attend all the study-associated visits.

Exclusion Criteria:

1. Patients who had received radiation therapy to the head and neck region.
2. Patients with other systemic diseases known to cause xerostomia (Sjogren's syndrome, rheumatoid arthritis, systemic lupus erythematosus, hepatitis C virus, tuberculosis, or sarcoidosis).
3. Patients using any other medication for their dry mouth condition (pilocarpine, cevimeline) 7 days before entering into the study.
4. Patients requiring hospitalization for any medical problem during the study.
5. Known hypersensitivity to the active ingredient of the product that will be used as assessed by the medical history questionnaire.
6. Vulnerable groups such as mentally or physically handicapped individuals, pregnant females, prisoners.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change in unstimulated Salivary flow rate | Baseline, 2weeks and 4weeks
  Milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Radwa Rageb, PHD, Study Director — Ain Shams University
Locations (1):
- Faculty of dentistry Ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No